CLINICAL TRIAL: NCT04381624
Title: Transcutaneous Vagal Stimulation in Knee Osteoarthritis (TRAVKO): Protocol of a Superiority, Outcome Assessor- and Participant-blind, Randomised Controlled Trial.
Brief Title: Transcutaneous Vagal Stimulation in Knee Osteoarthritis
Acronym: TRAVKO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universidad de La Frontera (Other)
Responsible Party: Principal Investigator, Germán Gálvez García, PhD, Universidad de La Frontera
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FONIS SA19/0003
Record Dates: First submitted 2020-04-18; First posted 2020-05-11 (Actual); Last update posted 2022-12-13 (Actual); Status verified 2022-12

CONDITIONS: Osteoarthritis, Knee
Keywords: pain; pain management; transcutaneous vagal stimulation; exercise
MeSH Terms: conditions — Osteoarthritis, Knee; Pain; Agnosia; Motor Activity | interventions — Resistance Training

STUDY DESIGN:
Intervention Model Description: randomised controlled, two-arm, double-blind
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transcutaneous Vagal Stimulation (Experimental): TVS will be applied through a portable electrostimulation equipment during the whole session in each of the treatment sessions. The electrodes will be placed in the left ear, specifically in the auricular concha. The device will be programmed with a biphasic square current at an intensity that produces a clear tingling sensation that is neither uncomfortable nor painful, with pulses of 300 microseconds, at 25 Hertz, the stimulus will be present for 30 seconds and will be followed by a 30-second rest period repeating this for approximately one hour.
  Interventions: Other: Exercise program
- Sham Transcutaneous Vagal Stimulation (Placebo Comparator): The device will be configured with the same parameters and intensity of the real TVS. However the device will be located in the left ear lobe.
  Interventions: Other: Exercise program

INTERVENTIONS:
Other: Exercise program — exercise program in 12 sessions, of approximately one hour, distributed in 3 sessions per week during a month

SUMMARY:
This study will evaluate the efficacy of Transcutaneous Vagal Stimulation in people whit knee osteoarthritis.

DETAILED DESCRIPTION:
Current treatments for knee osteoarthritis (KOA) are partially effective. It is, therefore, necessary to find new strategies that can complement the existing ones. In this scenario, transcutaneous vagal stimulation (TVS) neurophysiological effects could be a helpful solution. However, there is no evidence of the efficacy of TVS in KOA. This trial aims to assess the efficacy of TVS in decreasing pain in participants aged 55 years or older with KOA. A randomised controlled, two-arm, double-blind (participants and outcome assessors) and clinical superiority trial will be conducted for 70 patients with KOA. All the participants will carry out an exercise program. It consists of 12 sessions over four weeks. In addition, they will be randomly assigned to (1) active TVS plus physical exercise or (2) sham TVS plus physical exercise. The application of active TVS consists of electronic stimulation of the auricular concha using a portable device. Sham TVS condition consists of the stimulation of the earlobe that does not cause neurophysiological effects. The primary outcome is the reduction in pain intensity. Additionally, functional capacity, physical performance, pain-related interference, pain-related distress, quality of life in older adults and global change will be measured. Assessments will be conducted at the beginning of the study (baseline), at the end of the intervention and after 1 and 3 months of follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Women and men aged 55 and over;
2. Medical diagnosis of osteoarthritis of the knee according to the criteria of the American College of Rheumatologists;
3. Chronic pain (i.e., 3 months or more)
4. Average pain of the last seven days among 30 mm and 80 mm on the Visual Analogue Scale;
5. Walking without technical aids or knee brace;
6. Availability to attend an exercise program three times a week for four weeks;
7. Access to communication via telephone;
8. Agree to participate in the study by signing an informed consent form.

Exclusion Criteria:

1. Presence of the following symptoms and signs: Fever or chills, large effusions, paresthesias or paresis of the lower limb;
2. Presence of medically diagnosed psychiatric or neurological diseases (cognitive impairment, Alzheimer's, Parkinson's, epilepsy, moderate or severe depression, bipolar disorders, obsessive-compulsive disorder, etc.)
3. Neuromuscular or cardiac disorders (i.e., arrhythmia, conduction cardiac block), stroke, generalised rheumatology, dia-betes mellitus II, morbid obesity (i.e., equal to or greater than III);
4. Medical contraindication of physical exercise;
5. Joint infiltration or lower limb surgery in the previous 6 months;
6. Surgery is planned for the next 6 months;
7. Take strong regular two or more kinds of medication;
8. Conditions that affect the lower limb and/or limit its functional capacity, such as previous fractures in the area, deformity, joint replacement, tibial osteotomy;
9. Participation in exercise programs in the last nine months;
10. Inability to follow instructions.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2023-03-01 (Estimated); Primary Completion 2023-12-25 (Estimated); Study Completion 2024-03-01 (Estimated)

PRIMARY OUTCOMES:
average of the last seven days (VAS-7D) | at the end of treatment (1 month), 1 month, and 3 months of follow-up
  It will be evaluated through the Visual Analog Scale (VAS). This consists of a 100 mm horizontal line. On the left extreme it says "no pain" and on the right extreme decree it says "worst pain imaginable". The individual must indicate the intensity of pain by means of a mark. The result will be expressed by millimetres.

SECONDARY OUTCOMES:
intensity of the pain at rest (VAS-R) and walking on flat ground (VAS-W) | Baseline, at the end of treatment (1 month), 1 month, and 3 months of follow-up
  It will be evaluated through the Visual Analog Scale (VAS). This consists of a 100 mm horizontal line. On the left extreme it says "no pain" and on the right extreme decree it says "worst pain imaginable". The individual must indicate the intensity of pain by means of a mark. The result will be expressed by millimetres.
Functional capacity | Baseline, at the end of treatment (1 month), 1 month, and 3 months of follow-up
  Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC). The range of values is from 0 to 100. Lower values indicate greater functional capacity and vice versa.
Pain-related interference | Baseline, at the end of treatment (1 month), 1 month, and 3 months of follow-up
  How pain interferes with the individual's daily activities is described (Treede et al., 2019). It will be assessed through an VAS that on its left end will locate the absence of interference (ie, "no interference") and on its right end will locate the maximum interference (ie, "unable to perform my activities")
Pain-related distress | Baseline, at the end of treatment (1 month), 1 month, and 3 months of follow-up
  Unpleasant multifactorial emotional experience of a psychological (cognitive, behavioral and emotional), social or spiritual nature, due to persistent or recurring pain. It will be assessed by asking the participant to rate the pain-related distress they experienced in the past week on an VAS that will locate the absence of distress on its left end (ie, "no pain related distress") and on its right end will locate the maximum intensity of distress (ie, "Extreme distress related to pain")
Quality of life in older adults | Baseline, at the end of treatment (1 month), 1 month, and 3 months of follow-up
  It will be measured with WHOQOL-BREF. It contains four dimensions from which scores are obtained separately. Scores range from 0 to 100. Higher scores indicate better quality of life.
Global change | at the end of treatment (1 month), 1 month, and 3 months of follow-up
  It will be evaluated with the Patient-perceived satisfactory improvement. These was constructed using a 5-point categorical rating of change scale (''worse'', ''unchanged'', ''unsatisfactory improved'', ''satisfactory improved'' and ''good to very good improved'')
Session attendance | at the end of treatment (1 month)
  physical therapist treatment notes
Adverse Events | at the end of treatment (1 month)
  Adverse Events will be recorded, which will be understood as the perception of any problem that the participant attributes to his or her participation in the study and which requires him or her to be absent from 2 or more sessions or to seek external treatment
Gait speed test | Baseline, at the end of treatment (1 month)
  Meters per second
Standing and sitting in 30 seconds | Baseline, at the end of treatment (1 month)
  Number of repetitions
Time up and go | Baseline, at the end of treatment (1 month)
  Seconds
Unipodal stance task | Baseline, at the end of treatment (1 month)
  Seconds

OTHER OUTCOMES:
Kinesiophobia | Baseline, at the end of treatment (1 month)
  It will be evaluated using the Kinesiophobia TAMPA Scale. It is expressed on a scale of 11 to 44 points, where the highest score is related to the highest level of kinesiophobia.
Sleep Quality | Baseline, at the end of treatment (1 month)
  Sleep quality will be measured through the Pittsburgh Sleep Quality Index (PSQI). Sleep quality score is express in a scale from 0 to 21 points, where the highest score is related with worst sleep quality.
Pain Catastrophism | Baseline, at the end of treatment (1 month)
  This will be evaluated using the Pain Catastrophism Scale. It is expressed on a scale of 0 to 52 points, where the highest score is related to the highest level of catastrophism.
Negative Affectivity | Baseline, at the end of treatment (1 month)
  This will be evaluated using Depression, Anxiety and Stress Scale - 21 (DASS-21). The scale is expressed as a score from 0 to 63 points. Higher score reflects greater negative affectivity.
Pain Self-Efficacy | Baseline, at the end of treatment (1 month)
  This will be evaluated using the Pain self-efficacy questionnaire. The scale is expressed from 0 to 60 points. Higher score reflects greater perception of self-efficacy.

CONTACTS AND LOCATIONS:
Overall Officials: Claudio Bascour, PhD, Principal Investigator — Universidad de La Frontera
Locations (1):
- Universidad de La Frontera, Temuco, La Araucania, Chile

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in the main results article, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol
Time Frame: Beginning 3 months following main results article publication
Access Criteria: Investigators whose proposed use of the data has been approved by an independent review committee ("learned intermediary") identified for this purpose.
  For individual participant data meta-analysis. Proposals should be directed to Principal Investigator. To gain access, data requestors will need to sign a data access agreement